CLINICAL TRIAL: NCT00798226
Title: Fish Oil Supplementation During Pregnancy for Prevention of Asthma, Eczema and Allergies in Childhood: Interventional Trial in the COPSAC2010 (Copenhagen Studies on Asthma in Childhood) Birth Cohort
Brief Title: Fish Oil Supplementation During Pregnancy for Prevention of Asthma, Eczema and Allergies in Childhood
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Copenhagen Studies on Asthma in Childhood (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-B-2008-093
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Asthma; Eczema; Allergy
Keywords: Asthma; Eczema; Sensitization; Allergy
MeSH Terms: conditions — Asthma; Eczema; Hypersensitivity | interventions — Fatty Acids, Omega-3; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- 1 (Active Comparator): n-3 fatty acid
  Interventions: Dietary Supplement: n-3 fatty acid
- 2 (Placebo Comparator): Olive oil
  Interventions: Dietary Supplement: olive oil

INTERVENTIONS:
Dietary Supplement: n-3 fatty acid — Oral intake of 4 capsules daily from week 24 of gestation to 1 week after delivery
  Other Names: Incromega (Croda Nordica AB), Krossverksgatan 5 C, SE-216 16 Limhamn, Sweden
  Arms: 1
Dietary Supplement: olive oil — Oral intake of 4 capsules (1 g) daily from 24 weeks of gestation to 1 week after delivery
  Other Names: Pharmatech AS, Po 85, 1662 Rolvsøy, Norway
  Arms: 2

SUMMARY:
The aim of this study is to prevent asthma and allergies in childhood by supplementation with fish oil (n-3 fatty acids) to the mother during pregnancy. Paticipants are mother and children participating in the ABC-(Asthma Begins in Childhood)cohort. Mothers are recruited during pregnancy and receive supplement with n-3 fatty acids or olive oil (placebo) from week 24 of gestation to 1 week after delivery. The child is followed with acute and planned visit at the research unit and diagnosis of disease is done in the research unit according to predefined algorithms.

ELIGIBILITY:
Inclusion Criteria (mother):

* Pregnant women
* Living in Sealand, Denmark
* Fluent in Danish Language
* Willing to let the newborn child participate in the study

Exclusion Criteria (mother):

* Participating in other clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2008-11-26 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Persistent wheeze 0 to 3 years of age | 3 years
  Age at onset of persistent wheeze diagnosed according to predefined algorithm of recurrent troublesome lung symptoms, response to treatment and relapse after withdrawal of treatment

SECONDARY OUTCOMES:
Asthma exacerbations | 0-3 years
  Age at onset of severe asthma exacerbation diagnosed by predefined criteria of acute severe asthma requiring oral/high dose inhaled steroids or acute hospital contact
Infections | 0-3 years of age
  Main analysis:
  • Number of lower respiratory tract infections registered in daily diaries
  Secondary analyses:
  * Acute otitis media
  * Number of upper respiratory tract infections
  * Number of other infections
  * Total number of infections
Growth | 0 to 3 years of age
  * Body composition (fat mass and bone mineral density) assessed by DEXA scan at 3 years of age
  * Development of BMI from birth to 3 years assesses longitudinally in the research clinic
Neurological development | 0-3 years
  Main analysis:
  • Cognitive development assessed at 2½ years using the cognitive part of Bayley Scales of Infant and Toddler Development, third edition
  Secondary analyses:
  * Milestone development monitored prospectively by the parents using a registration form based on The Denver Development Index and WHO milestones registration (combined assessment by principal component analysis)
  * Language development assessed at 1 and 2 years of age with the Danish version of The MacArthur Bates Communicative Developmental Inventory (CDI)
  * The child´s general development (language, fine and gross motor, social and problem solving) at 3 years of age assessed with Ages and stages Questioner, third edition (ASQ-3)
Eczema | 0-3 years
  Age at onset of eczema diagnosed prospectively by research doctors according to predefined algorithm based upon Hanifin and Rajka criteria
Allergic sensitization | 6 and 18 months of age
  Allergic sensitization at 6 and/or 18 months of age assessed by skin prick test and specific IgE in blood
Systemic immune status | 18 months
  Main analysis
  * Immune status at 18 months measured in stimulated whole blood as cytokine release (combined assessments by prinicipal component analyses) Secondary analyses
  * Composition of immune cell subsets in whole blood at birth and at 18 months of age
Airway mucosal immune status | 4 weeks and 2 years of age
  Immune status measured in airway mucosal lining fluid at 4 weeks and 2 years of age (combined assessments by prinicipal component analyses for each age point)

OTHER OUTCOMES:
Asthma | 3-10 years of age
  Asthma diagnosed from age 3 to 10 years based on the same predefined algorithm of recurrent troublesome lung symptoms, response to treatment after withdrawal of treatment, which was used for persistent wheeze at age 0-3 in phase 1 of the study. Primary outcome in phase 2 is current asthma at specific visits till age 10 years, which is diagnosed in children fulfilling the persistent wheeze algorithm at any point during the first 10 years of life and still needing inhaled corticosteroids at specific visits (3, 4, 5, 6, 8 and 10 years of age) to control the symptoms.
Infections | 3-10 years of age
  Prescribed medicine for infections. Types and length of infections
Weight | 3-10 years of age
  Clinical follow up on the development of weight in kg (calibrated digital weight scales) at every visit till age 10 years assessed longitudinally in the research clinic.
Behavioral and psychopathological dimensions. | 10 years of age
  Behavioral and psychopathological dimensions will be assessed at 10 years of age.
  The childrens' potential psychiatric diagnoses will be ascertained through the semi-structured clinical interview Schedule for Affective Disorders and Schizophrenia for School-Age Children - Present and Lifetime Version (K-SADS-PL) first with a parent and next with the child.
MRI scanning of the brain | 10 years of age
  MRI scanning of the brain. The scanning procedure will take up to 1 hour.
Eczema | 3-10 years of age
  Age at onset of eczema diagnosed prospectively by research doctors according to predefined algorithm based upon Hanifin and Rajka criteria.
Allergic sensitization/atopy | 6-10 years of age
  Allergic sensitization at 6 and 10 years of age assessed by skin prick test (ALK-Abelló, Denmark).
Airway mucosal immune status: | 3-10 years of age
  Immune status measured in airway mucosal lining fluid at 3, 6 and 10 years of age (combined assessments by principal component analyses for each age point).
Allergic rhinitis | 3-10 years of age
  Allergic rhinitis will be diagnosed by combining allergic sensitization with symptom recording of troublesome congestion or sneezing or runny nose upon relevant exposure to allergens at age 3, 4, 5, 6, 8 and 10 years.
Lung function measurements | [Time Frame: 5-10 years of age]
  Spirometry measuring airflow in liter. Compared with age and sex validated standards
Cognitive function | 10 years of age
  A 2,5 hours cognitive evaluation at 10 years of age. Cognitive functions from a broad spectrum of cognitive domains will be assessed with subtests both using paper pencil tests and Cambridge Neuropsychological Test Automated Battery .
Asthma exacerbations: | [Time Frame: 3-10 years of age]
  Age at onset and number of severe asthma exacerbation diagnosed by predefined criteria of acute severe asthma requiring oral/ high dose inhaled steroids or acute hospital contact
Body composition: | [Time Frame: 3-13 years of age]
  Body composition measured as fat mass, lean mass, bone mineral content (BMC) and bone mineral density assessed (BMD) through DXA scans at 3, 6 and 13 years of age.
  Body impedance measurements at 10 years of age.
Airway resistance | [Time Frame: 3-10 years of age]
  sRaw measured by plethysmography at age 3, 4, 5, 6, 8 and 10 years.
Airway resistance | [Time Frame: 3-5 years of age]
  Multiple breath wash-out using SF6 and N2 as inert gasses to determined LCI, Scond and Sacin at ages 3, 4 and 5 years.
Bronchial reactivity: | 6 years of age.
  Provocative dose of methacholine leading to a 20% drop in FEV1 from baseline (PD20 value) at age 6 years.
Airway inflammation: | [Time Frame: 6-10 years of age]
  Measurement of fractional exhaled nitric oxide (FeNO) at age 6, 8 and 10 years
Height | [Time Frame: 3-10 years of age]
  Clinical follow up on the development of height in cm (Harpenden stadiometer) at every visit till age 10 years assessed longitudinally in the research clinic.
Waistcircumference | [Time Frame: 3-10 years of age]
  Clinical follow up on the development of waistcircumference in cm(using tape; 3 times each) at every visit till age 10 years assessed longitudinally in the research clinic.
Headcircumference | [Time Frame: 3-10 years of age]
  Clinical follow up on the development of headcircumference in cm(using tape; 3 times each) at every visit till age 10 years assessed longitudinally in the research clinic.
Thoraxcircumference | [Time Frame: 3-10 years of age]
  Clinical follow up on the development of thoraxcircumference in cm(using tape; 3 times each) at every visit till age 10 years assessed longitudinally in the research clinic.
Strength and Difficulties Questionnaire (SDQ)- Questionnaires | 6, 8 and 10 years of age.
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire about 3-16 year olds. Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology and behavior problems. Scores will be calculated form the questionnaires in order validated methods
ADHD- RS- Questionnaires | 8 and 10 years of age.
  The ADHD Rating Scale obtains parent ratings regarding the frequency of each ADHD symptom based on DSM criteria.
  Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology and behavior problems. Scores will be calculated form the questionnaires. Scores will be calculated form the questionnaires in order validated methods.
Social Responsive Scale, Second version (SRS-2) | 10 years of age
  The SRS-2 identifies social impairment associated with autism spectrum disorders (ASDs) and quantifies its severity Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology. Scores will be calculated form the questionnaires. Scores will be calculated form the questionnaires in order validated methods.
The Behavior Rating Inventory of Executive Function 2nd edition (BRIEF-2) | 10 years of age
  The BRIEF-2 is a set of questionnaires for parents and teachers , designed to evaluate executive function from multiple perspectives.
  Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology. Scores will be calculated form the questionnaires. Scores will be calculated form the questionnaires in order validated methods.
The Child Behavior Checklist school-age version (CBCL) | 10 years of age
  The Child Behavior Checklist (CBCL) is a widely used questionnaire to assess behavioral and emotional problems.
  Questionnaires will be administered to the parents to obtain their evaluation of their child's potential psychopathology and behavior problems. Scores will be calculated form the questionnaires. Scores will be calculated form the questionnaires in order validated methods.
Allergic sensitization | 6 and 10 years of age
  Allergic sensitization assessed specific IgE in blood (ImmunoCAP, PHarmacia Diagnostics AB, Sweden).

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Bønnelykke, MD, PhD, Principal Investigator — COPSAC / University of Copenhagen
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital of Copenhagen, Gentofte Municipality, Gentofte
  - Næstved Hospital, Pediatric Department, Næstved, Næstved

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen L, Brustad N, Luo Y, Wang T, Ali M, Ebrahimi P, Schoos AM, Vahman N, Lovric M, Rasmussen MA, Kolmert J, Wheelock CE, Lasky-Su JA, Stokholm J, Bonnelykke K, Chawes B. Prenatal Fish Oil Supplementation, Maternal COX1 Genotype, and Childhood Atopic Dermatitis: A Secondary Analysis of a Randomized Clinical Trial. JAMA Dermatol. 2024 Oct 1;160(10):1082-1090. doi: 10.1001/jamadermatol.2024.2849. PMID 39196551
- [Derived] Vinding RK, Sevelsted A, Horner D, Vahman N, Lauritzen L, Hagen CP, Chawes B, Stokholm J, Bonnelykke K. Fish oil supplementation during pregnancy, anthropometrics, and metabolic health at age ten: A randomized clinical trial. Am J Clin Nutr. 2024 Apr;119(4):960-968. doi: 10.1016/j.ajcnut.2023.12.015. Epub 2024 Feb 22. PMID 38569788
- [Derived] Bisgaard H, Mikkelsen M, Rasmussen MA, Sevelsted A, Schoos AM, Brustad N, Eliasen AU, Thorsen J, Chawes B, Gurdeniz G, Morin A, Stark K, Stokholm J, Ober C, Pedersen CET, Bonnelykke K. Atopic and non-atopic effects of fish oil supplementation during pregnancy. Thorax. 2023 Dec;78(12):1168-1174. doi: 10.1136/thorax-2022-219725. Epub 2023 Sep 11. PMID 37696621
- [Derived] Prince N, Kelly RS, Chu SH, Kachroo P, Chen Y, Mendez KM, Begum S, Bisgaard H, Bonnelykke K, Kim M, Levy O, Litonjua AA, Wheelock CE, Weiss ST, Chawes BL, Lasky-Su JA. Elevated third trimester corticosteroid levels are associated with fewer offspring infections. Sci Rep. 2023 Jun 28;13(1):10461. doi: 10.1038/s41598-023-36535-0. PMID 37380711
- [Derived] Brustad N, Yang L, Chawes BL, Stokholm J, Gurdeniz G, Bonnelykke K, Bisgaard H. Fish Oil and Vitamin D Supplementations in Pregnancy Protect Against Childhood Croup. J Allergy Clin Immunol Pract. 2023 Jan;11(1):315-321. doi: 10.1016/j.jaip.2022.09.027. Epub 2022 Sep 30. PMID 36184023
- [Derived] Horner D, Hjelmso MH, Thorsen J, Rasmussen M, Eliasen A, Vinding RK, Schoos AM, Brustad N, Sunde RB, Bonnelykke K, Chawes BL, Stokholm J, Bisgaard H. Supplementation With Fish Oil in Pregnancy Reduces Gastroenteritis in Early Childhood. J Infect Dis. 2023 Feb 1;227(3):448-456. doi: 10.1093/infdis/jiab607. PMID 34927195
- [Derived] Vinding RK, Stokholm J, Sevelsted A, Chawes BL, Bonnelykke K, Barman M, Jacobsson B, Bisgaard H. Fish Oil Supplementation in Pregnancy Increases Gestational Age, Size for Gestational Age, and Birth Weight in Infants: A Randomized Controlled Trial. J Nutr. 2019 Apr 1;149(4):628-634. doi: 10.1093/jn/nxy204. PMID 30418579
- [Derived] Vinding RK, Stokholm J, Sevelsted A, Sejersen T, Chawes BL, Bonnelykke K, Thorsen J, Howe LD, Krakauer M, Bisgaard H. Effect of fish oil supplementation in pregnancy on bone, lean, and fat mass at six years: randomised clinical trial. BMJ. 2018 Sep 4;362:k3312. doi: 10.1136/bmj.k3312. PMID 30181143
- [Derived] Bisgaard H, Stokholm J, Chawes BL, Vissing NH, Bjarnadottir E, Schoos AM, Wolsk HM, Pedersen TM, Vinding RK, Thorsteinsdottir S, Folsgaard NV, Fink NR, Thorsen J, Pedersen AG, Waage J, Rasmussen MA, Stark KD, Olsen SF, Bonnelykke K. Fish Oil-Derived Fatty Acids in Pregnancy and Wheeze and Asthma in Offspring. N Engl J Med. 2016 Dec 29;375(26):2530-9. doi: 10.1056/NEJMoa1503734. PMID 28029926